CLINICAL TRIAL: NCT05593471
Title: Influences of High Versus Low-intensity Exercises in Post-COVID-19 Patients With Sarcopenia Secondary to Chronic Kidney Disease: Randomized Controlled Trial
Brief Title: Low Versus High-intensity Exercises in Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, assistant professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCR-22029
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity exercises (Experimental): The first group (HG) received a High-intensity exercise program consisting of progressive resistance training for 30 min using dumbbells, sandbags, and TheraBand with different colors. The exercised muscles were (knee extensors, elbow flexors, chest muscles, hip adductors, abductors, abdominal muscles, back muscles, and hand grip muscles) (references). The intensity of exercise was determined by the load which was kept at 65% of the 10-repetition maximum throughout the program duration. The repetitions of each exercise were kept at a fixed value of 2 sets of 10 - 12 repetitions per session (exercises stopped if the patient reached fatigue level). For progression, the 10-repetition maximum test was performed on a weekly schedule and the amount of load was adjusted accordingly. Exercises were done in a cyclic manner where half of the selected muscles were exercised per session and the other half were exercised in the next session.
  Interventions: Other: high intensity exercises
- low intensity aerobic exercises (Experimental): The second group (LG) received a low-intensity aerobic exercise program consisting of an arm ergometer, and a bicycle ergometer to train both upper and lower body muscles. Additionally, 5 minutes of regular treadmill walking was added at the beginning and the end of the exercises session as warming up and cooling down respectively. Exercises were performed in a cyclic manner where the arm and bicycle ergometers were used alternatively. The rate of perceived exertion (RPE) scale was used to monitor the intensity of the exercises to be at 3 -4 level. The actual working out time was 20 minutes plus 10 minutes for the warming up and cooling down. Sessions were performed 3 times per week for six weeks.
  Interventions: Other: low intensity aerobic exercises

INTERVENTIONS:
Other: high intensity exercises — resistance training progressively increasing according to specific criteria (10 repetitions maximum). for the major muscles of the body
  Other Names: progressive resistance training
  Arms: High intensity exercises
Other: low intensity aerobic exercises — low-intensity exercises performed using arm or leg ergometer machines
  Other Names: aerobic exercises
  Arms: low intensity aerobic exercises

SUMMARY:
this study aims to compare the effect of high-intensity resistance exercises measured using the 10-repetition maximum versus low-intensity aerobic exercises on muscle performance, physical function and quality of life in chronic kidney patients with sarcopenia who recently recovered from COVID-19 infection

DETAILED DESCRIPTION:
Sarcopenia is a prevalent chronic disease caused by aging and is characterized by a reduction in muscle strength and mass (Barajas-Galindo et al., 2021), and consequently deterioration in physical function and quality of life (Gil et al., 2021; Tsekoura et al., 2017). Sarcopenia is associated with higher rates of stroke, frailty, (Bikbov et al., 2020; Go et al., 2004; Levin et al., 2013), and mortality (Ali & Kunugi, 2021). Generally, there are numerous causes of sarcopenia, including chronic kidney diseases (CKD) (Souza et al., 2017), environmental factors, inflammatory mediator's activation, physical inactivity, mitochondrial dysfunction, hormonal changes, and loss of neural junctions (Walston, 2012).

Recently, Sarcopenia had great attention, especially among patients with CKD who already suffer from increased catabolism, higher protein wasting, and other metabolic disorders and decreased functional reserve. Additionality, the decline in physical function due to the deterioration of muscle mass, power, and strength could significantly decrease balance and increase the risk of falling in these populations (Moorthi & Avin, 2017).

After the pandemic of COVID-19 and the mandatory quarantine of patients during the recovery period, CKD patients with sarcopenia who were infected with COVID-19 will be forced to assume a more sedentary lifestyle which consequently magnifies all health risks (Gérard et al., 2021; Gil et al., 2021) jeopardize subjects vitality (Morley et al., 2020; Mousa et al., 2021) and increasing prevalence of sarcopenia (Ali & Kunugi, 2021).

Exercise has been proposed as one of the solutions for sarcopenia-associated symptoms. As per a recent systematic review (Barajas-Galindo et al., 2021), resistance exercises alone or with other forms of exercises could be beneficial especially in improving anthropometric parameters and muscle performance. Yet its specific effects on post-COVID-19 CKD patients who have sarcopenia need further investigation.

The aim of this study is to compare the effectiveness of high versus low-intensity exercises on muscle strength, and physical function in post-COVID-19 patients with sarcopenia secondary to CKD.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes with age between 50 - 70 years old.
* CKD stages (3 and 4)
* Infected by COVID-19 and recovered (1 - 2 months)
* Score of 4 or more on SAR-QoL Questionnaire
* Patients having had a medical prescription for physical rehabilitation.

Exclusion Criteria:

* Patients infected again by -CoVID-19
* Any serious inflammatory, neurological, or cardiovascular diseases.
* Chronic chest disease.
* Chronic inflammatory orthopedic disorders and rheumatoid arthritis.
* Mental impairments.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Quality of life (SAR QoL) questionnaire used to assess the quality of life experienced by sarcopenia patients | 6 weeks
  In order to measure the quality of life, we used the SarQoL® questionnaire, which is a valid, consistent, and reliable, and can therefore be recommended for clinical and research purposes (Beaudart et al., 2017).

SECONDARY OUTCOMES:
Physical function: | 6 weeks
  Modified Physical Performance Test (MPPT) was used to assess basic and complex functional abilities Activities of Daily Living (ADL) with varying difficulty levels. During the test, nine standardized tasks are performed (including walking 15.2 meters, doing a 360° turn, putting on a coat, picking up a coin, rising from a chair, lifting a book, climbing stairs in 2 variations, and picking up a coin). (Brown et al., 2000)
Muscle power: | 6 weeks
  (STS- 60): Muscle physical performance is better represented by STS tests than muscle strength. The test used determines which subsets of the population are at risk for sarcopenia. This test measures patient exercise capacity and leg muscle strength. As fast as patient can within a minute, stand up from the chair with his legs straight and sit back down (Bohannon & Crouch, 2019; Yee et al., 2021)
Muscle strength | 6 weeks
  isometric hand-grip strength was performed using the JAMAR hand dynamometer (Sammons Preston Rolyan, Bolingbrook, Illinois) were used to measure hand-grip strength of the dominant hand. The participants were seated with their elbows flexed at 90° and their trunks resting. Individual grip sizes were adjusted. Two attempts were conducted, and the averaged values was recorded (Huang et al., 2022; Stoever et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid Hospital, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No